CLINICAL TRIAL: NCT03869827
Title: Evaluation of the Risk of Necrotizing Enterocolitis in Fetuses With Intrauterine Growth Restriction.
Brief Title: Necrotizing Enterocolitis in Fetuses With Intrauterine Growth Restriction
Acronym: ECUN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: ECUN
Record Dates: First submitted 2019-03-04; First posted 2019-03-11 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IUGR: All birth between 24 + 0 weeks of amenorrhea and 36 + 6 weeks of amenorrhea with isolated intrauterine growth restriction at the maternity ward of the hospital Femme-Mère-Enfant from 1st of january 2011 to 31 december 2016.
  Interventions: Other: necrotizing enterocolitis
- Control: To each of these children with intrauterine growth restriction is matched a control child: the child without intrauterine growth restriction of the same gestational age whose date of birth is consecutive to that of the case.
  Interventions: Other: necrotizing enterocolitis

INTERVENTIONS:
Other: necrotizing enterocolitis — Collection of necrotizing enterocolitis diagnosis, as well as its severity, are based on the classification of Belle modified in 3 stages: 1) Suspected, 2) Proven, 3) Advanced

SUMMARY:
Necrotizing enterocolitis is the most common gastroenterological emergency in neonatology. Its mortality is high, ranging from 15 to 30%. Prematurity is the main risk factor for necrotizing enterocolitis, as well as the very low birth weight (<1500 g) associated with prematurity. Among the early neonatal complications of intrauterine growth restriction neonates, necrotizing enterocolitis is frequently reported in the literature. The situation of chronic hypoxia of these fetuses is at the origin of a vascular redistribution favoring the cerebral circulation to the detriment of the mesenteric vascularization, which could lead to the development of an necrotizing enterocolitis. However, data from the literature concerning this over-risk of necrotizing enterocolitis in the case of intrauterine growth restriction are discordant. The heterogeneity of the definitions used for the intrauterine growth restriction and diagnostic criteria for necrotizing enterocolitis from one study to another could explain these discrepancies. The investigator's hypothesis is that the risk of necrotizing enterocolitis is higher among newborns in intrauterine growth restriction compared to control children.

ELIGIBILITY:
Inclusion Criteria:

* All birth between 24 + 0 weeks of amenorrhea and 36 + 6 weeks of amenorrhea
* with isolated intrauterine growth restriction at the maternity ward of the hospital Femme-Mère-Enfant
* from 1st of january 2011 to 31 december 2016.

Inclusion Criteria for control group:

* All birth between 24 + 0 weeks of amenorrhea and 36 + 6 weeks of amenorrhea
* without isolated intrauterine growth restriction at the maternity ward of the hospital Femme-Mère-Enfant
* from 1st of january 2011 to 31 december 2016.

Exclusion Criteria:

* Infants born out of the hospital and secondarily hospitalized in our department
* unaccompanied pregnancies
* multiple pregnancies
* children with malformations or genetic abnormalities,
* medical termination of pregnancy
* fetal deaths in utero

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All birth between 24 + 0 weeks of amenorrhea and 36 + 6 weeks of amenorrhea with isolated intrauterine growth restriction at the maternity ward of the hospital Femme-Mère-Enfant from 1st of january 2011 to 31 december 2016.
  To each of these children with intrauterine growth restriction is matched a control child: the child without intrauterine growth restriction of the same gestational age whose date of birth is consecutive to that of the case.
Sampling Method: Non-Probability Sample
Enrollment: 378 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Necrotizing Enterocolitis stage 1 | between 2011 and 2016
  The necrotizing enterocolitis diagnosis, as well as its severity, are based on the classification of Belle modified in 3 stages: 1) Suspected, 2) Proven, 3) Advanced
Number of patients with Necrotizing Enterocolitis stage 2 | between 2011 and 2016
  The necrotizing enterocolitis diagnosis, as well as its severity, are based on the classification of Belle modified in 3 stages: 1) Suspected, 2) Proven, 3) Advanced
Number of patients with Necrotizing Enterocolitis stage 3 | between 2011 and 2016
  The necrotizing enterocolitis diagnosis, as well as its severity, are based on the classification of Belle modified in 3 stages: 1) Suspected, 2) Proven, 3) Advanced

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Doret, ¨Prof., Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France